CLINICAL TRIAL: NCT05666843
Title: The Effects of Personalized Dietary Guidance to Increase the Intake of Fibre-rich Foods on Cardiometabolic Risk Profile in Individuals With Type 2 Diabetes. (in Dutch: Voed je Beter Met Diabetes Type 2)
Brief Title: Dietary Intervention to Improve Cardiometabolic Risk Profile in Individuals With Type 2 Diabetes
Acronym: VJBD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Marianne Geleijnse, prof.dr. JM (Marianne) Geleijnse, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL80697.091.22
Record Dates: First submitted 2022-11-17; First posted 2022-12-28 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: dietary guidelines; dietitian; dietary fiber; diabetes type 2; nutrition; randomized controlled trial (RCT); cardiovascular diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The nature of the intervention does not allow for blinding of the participants or researchers. After data collection, the database will be coded by an independent researcher to ensure that data analysis is conducted in a blinded way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Personalized dietary guidance to increase the intake of fibre-rich foods on top of usual care. The dietary guidance is implemented by dieticians and is personalized based on current adherence to the dietary guidelines, usual dietary intake, gender and personal goals and preferences.
  Interventions: Behavioral: Personalized Dietary Advice
- Usual care group (No Intervention): Participants in the control group receive usual health care as provided by general practitioners and nurse practitioners or other health care professionals involved in diabetes care.

INTERVENTIONS:
Behavioral: Personalized Dietary Advice — Personalized dietary guidance to increase the intake of fibre-rich foods on top of usual care.The dietary guidance is implemented by dieticians and is personalized based on current adherence to the dietary guidelines, usual dietary intake, gender and personal goals and preferences.
  Arms: Intervention group

SUMMARY:
This is a randomized controlled trial to examine whether personalized guidance to increase the consumption of fiber rich food items according to the Dutch dietary guidelines, compared to usual care, improves health of individuals with type 2 diabetes.

DETAILED DESCRIPTION:
Previous interventions with fibre supplements show promising results among individuals with type 2 diabetes, but wether these effects are similar when higher fiber intake is achieved through diet and not through supplements remains unclear.

The primary objective of this study is to investigate the effects of personalized dietary guidance to increase the intake of fibre-rich foods, as recommended in the Dutch dietary guidelines, on cardiometabolic risk profile in individuals who have type 2 diabetes, compared to usual care after six months.

The study is a parallel randomized trial over a period of twelve months, including an intervention period of six months and a follow up period of six months. The study population consists of adults with non-insulin-dependent type 2 diabetes, diagnosed by a medical doctor at least 6 months prior to study enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes made by a medical doctor at least 6 months prior to study enrolment
* Adult
* Willing and able to follow dietary intervention
* Willing to participate in both intervention and control group
* Living at a reasonable distance from the research center at Wageningen University & Research (WUR) (i.e.maximum of ± 1 hour away)

Exclusion Criteria:

* Currently treated with insulin therapy
* Recently (< 6 months) or currently being under supervision of a dietician
* Pregnant or breast-feeding
* History of bariatric surgery, including gastric banding
* Current participation in a study with an investigational drug or dietary intervention
* Excessive alcohol consumption (more than 14 units for males/7 units for females per week) or drug use
* Clinical disorders that could interfere with the intervention (e.g. gastro-intestinal disorders, auto-immune diseases, psychiatric disorders, uncontrolled heart diseases, serious neurological disorders, renal failure or cancer)
* Not able to speak and understand the Dutch language
* No general practitioner
* Working at the department of Human Nutrition and Health at Wageningen University & Research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiometabolic risk profile (DIAL risk score) | Change from baseline at 6 months
  The change in cardiovascular risk based on observed changes in HbA1c, LDL-cholesterol and systolic blood pressure. DIAL risk score ranges from 0 to 100%, with higher scores indicating a higher risk.

SECONDARY OUTCOMES:
Cardiometabolic risk profile (DIAL risk score) | Change from baseline at 12 months
  The change in cardiovascular risk based on observed changes in HbA1c, LDL-cholesterol and systolic blood pressure. DIAL risk score ranges from 0 to 100%, with higher scores indicating a higher risk.
Body weight (in kilograms) | baseline, 6 months, 12 months
  As measured with a digital scale
Body mass index (kg/m^2) | baseline, 6 months, 12 months
  Weight and height will be combined to report BMI in kg/m^2.
Waist circumference | baseline, 6 months, 12 months
  in centimeters
Blood lipids | baseline, 6 months, 12 months
  Total cholesterol, HDL-cholesterol, LDL-cholesterol, Triglycerides
Dietary intake | baseline, 3 months, 6 months, 12 months
  Nutrient intake and diet quality score for the level of adherence to the Dutch dietary guidelines. Diet quality score (Dutch Healthy Diet index) ranges from 0-160, with higher scores indicating better diet quality.
Micronutrient status | baseline, 6 months, 12 months
  Micronutrient status as measured with biomarkers in blood and (24-hour) urine samples
Food literacy | baseline, 3 months, 6 months, 12 months
  Food literacy level by means of the 29-item Self Perceived Food Literacy Scale (SPFL-29). Scores range from 29-145, with higher scores indicating a higher level food literacy.
HbA1c | baseline, 6 months, 12 month
  As determined in blood samples
Fasting glucose | baseline, 6 months, 12 month
  As determined in blood samples
Fasting insulin | baseline, 6 months, 12 month
  As determined in blood samples
C-peptide | baseline, 6 months, 12 month
  As determined in blood samples
Blood pressure | baseline, 6 months, 12 months
  Systolic and diastolic blood pressure (mmHg) as determined with a digital blood pressure monitor
Estimated Glomerular Filtration Rate (eGFR) | baseline, 6 months, 12 months
  in ml/min/1,73 m2 as determined from blood sample
Urinary albumin levels | baseline, 6 months, 12 months
  in grams per deciliter (g/dL) as determined from urine sample
Liver function | baseline, 6 months, 12 months
  Aspartate transaminase (AST) and Alanine transaminase (ALT) ratio as determined from blood sample
Inflammatory markers | baseline, 6 months, 12 months
  hsCRP in blood samples
Quality of life score | baseline, 3 months, 6 months, 12 months
  Health related quality of life assessed with the 36-Item Short Form Survey (SF-36). Scores range from 0-100, with higher scores indicating higher quality of life.
Health index score | baseline, 3 months, 6 months, 12 months
  5-level EuroQol-5D version (EQ-5D). The maximum score of 1 indicates the best health state. In addition, there is a visual analogue scale (VAS) to indicate the general health status with 100 indicating the best health status.
Positive health score | baseline, 3 months, 6 months, 12 months
  Positive health is assessed with the 17-item Positive Health measurement scale. scores range from 0-170 with higher scores indicating higher positive health.
Self efficacy score | baseline, 3 months, 6 months, 12 months
  Self-efficacy as assessed with the Dutch General Self-Efficacy scale (DGSES). The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Sleep quality score | baseline, 3 months, 6 months, 12 months
  Sleep quality by means of Pittsburgh Sleep Quality Index (PSQI). A range of 0-21; higher scores indicate worse sleep quality.
Medical consumption | baseline, 3 months, 6 months, 12 months
  Medical consumption (incl. medication) by means of Institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ)
Productivity | baseline, 3 months, 6 months, 12 months
  Productivity by means of Institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (iPCQ)
Cardiovascular condition | baseline, 6 months, 12 months
  Heart rate (bpm) 1 minute after 3-minute step test
Leg muscle strength | baseline, 6 months, 12 months
  Measured as time to perform the 5 times sit-to-stand test (sec)
Balance score | baseline, 6 months, 12 months
  Tandem Romberg test score, range 0-4 with higher scores indicating better balance
Flexibility | baseline, 6 months, 12 months
  Measured as distance between finger and toes when performing the chair sit-and-reach test (cm)
Hand grip strength | baseline, 6 months, 12 months
  Hand grip strength (kg) using a hand-held dynamometer
Skeletal muscle fat infiltration | baseline, 6 months, 12 months
  Echo intensity of the skeletal muscle rectus femoris (ultrasound)

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Veldhuisen ER, van Damme I, Polhuis KCMM, Geleijnse JM, Winkels RM. The impact of a 6-month dietary counseling intervention on quality of life in individuals with type 2 diabetes: A secondary analysis of a randomized controlled trial. Clin Nutr ESPEN. 2025 Nov 22:102826. doi: 10.1016/j.clnesp.2025.11.146. Online ahead of print. PMID 41276175